CLINICAL TRIAL: NCT01027468
Title: Functional, Morphological And Safety Results After Intravitreal Bevacizumab Treatment Of Neovascular Age-related Macular Degeneration - 3 Years Of Follow-up
Brief Title: Long-term Results After Intravitreal Bevacizumab Treatment Of Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 548/2009
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: bevacizumab, choroidal neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Bevacizumab; Injections, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 1 (Experimental): bevacizumab intravitreal injection
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — intraocular bevacizumab injection
  Other Names: intraocular injection

SUMMARY:
200 eyes with each subtype of neovascular age-related macular degeneration will be included in this study and 3 years after the initial intravitreal bevacizumab, best-corrected visual acuity (BCVA) will be measured using Snellen charts at 6m. Central retinal thickness (CRT) will be measured using Stratus OCT and Cirrus SD-OCT (Zeiss). Data of treatment-naive eyes (group 1) were compared to the data of eyes that had undergone prior treatment with photodynamic therapy with verteporfin and intravitreal triamcinolone acetonide (group 2).

DETAILED DESCRIPTION:
In this interventional clinical study, 181 eyes of 160 consecutive patients with active neovascular related macular degeneration meeting recommended criteria for inclusion and protocol criteria for anti-vascular endothelial growth factor therapy undergoing intravitreal bevacizumab monotherapy were evaluated. Data of treatment-naive eyes (Group 1, n = 114) were analyzed separately from eyes that had undergone previous photodynamic therapy plus intravitreal triamcinolone (Group 2, n = 67). Re-treatment criteria were based on clinical outcome following the official European label regimen. After 1 year of continuous service at an academic referral center, follow-up was performed in private practices in collaboration with the referral center. Main outcome parameters were best-corrected visual acuity and central retinal thickness.

ELIGIBILITY:
Inclusion Criteria:

* any subtype of neovascular age-related macular degeneration
* age of 50 years or older
* initial treatment with intravitreal bevacizumab between August 2005 and June 2006

Exclusion Criteria:

* previous vitrectomy
* presence of cystoid macular edema without choroidal neovascularization
* Uncontrolled systemic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, PD Dr., Principal Investigator — Department of Ophthalmology, Medical University of Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical University of Vienna, Department of Ophthalmology during September 2008-July 2009 with a mean of 3 year follow-up after initial Bevacizumab intravitreal treatment
Pre-assignment Details: Inclusion criteria:
  * patients treated with bevacizumab due to wet age-related macular degeneration
  * follow-up of 3 years
  Exclusion criteria:
  - patients with other macular diseases
Groups:
- Group 1: 3 year follow-up of patients with intravitreal application of bevacizumab: From August 2005 to July 2006: 1 mg (0.04 mL) of bevacizumab After July 2006: 2.5 mg (0.1 mL) of Bevacizumab Follow-up intervals: 6-8 weeks
Period: Overall Study
Arm/Group | Group 1
Started | 160
Completed | 160
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: 3 year follow-up of intravitreal application of bevacizumab
Arm/Group | Group 1
Number analyzed (Participants) | 160
Age, Customized [Mean (Standard Deviation); unit: years] | 77.24 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Vision
Description: Best-corrected visual acuity converted to logMAR (MAR=minimum angle of resolution) for statistical analysis
Time Frame: 3 years after first intravitreal bevacizumab treatment
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Group 1
Number analyzed (Participants) | 160
logMAR | 0.16 (0.21)

2. Primary Outcome: CRT (Central Retinal Thickness)
Description: Central retinal thickness measured in µm
Time Frame: 3 years after initial intravitreal bevacizumab treatment
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Group 1
Number analyzed (Participants) | 160
µm | 319 (110)

3. Secondary Outcome: Systemic Complications After Treatment
Time Frame: 3 years after initial bevacizumab treatment
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 160
participants
  Retinal Detachment | 0
  Endophthalmitis | 0
  Severe intraocular inflammation | 5
  thromboembolic disease with myocardial infarction | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 5/160
Other Adverse Events (participants affected / at risk) | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=160)
intraocular inflammation (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes